CLINICAL TRIAL: NCT02711501
Title: Comparison of Post-operative Complications of Bone Augmentation at Anterior of Maxilla After Periosteal Releasing Incision With Two Techniques Diode Laser and Scalpel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Neda Moslemi, Associate Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TehranUMS h4p62mb2
Record Dates: First submitted 2016-02-04; First posted 2016-03-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Post-operative Pain
Keywords: post-operative pain; diode laser
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser irradiation (Experimental): laser-assisted surgery with the following parameters: Wavelength:810 nanometer, power: 3 W, pulse mode,pulse length 100 µs, pulse interval 200 µs
  Interventions: Procedure: Laser-assisted surgery.
- blade (Experimental): conventional surgery by blade
  Interventions: Procedure: conventional surgery by blade

INTERVENTIONS:
Procedure: Laser-assisted surgery. — laser-assisted surgery
  Arms: Laser irradiation
Procedure: conventional surgery by blade — conventional surgery
  Arms: blade

SUMMARY:
The aim of this study was to investigate if using lasers instead of scalpel for flap advancement in bone augmentation procedures would reduce post-operative swelling and pain.

DETAILED DESCRIPTION:
Guided bone regeneration (GBR) is a well established method to augment excessive alveolar bone loss before and at the time of implant placement. Primary closure of soft tissue is a prerequisite for successful bone augmentation procedures. Adequate flap advancement is a key factor for tension free primary wound closure. The tension free flap is usually attained by incising the buccal flap using scalpels. However, this procedure, especially in cases with major flap advancement, results in increased patient morbidity after surgery. Swelling and hemorrhage during the first week after surgery have a negative effect on patient's quality of life.

Currently, lasers are widely used as a tool for soft tissue management and diode laser appears to be an effective tool for incision and excision of the soft tissue. The major advantageous property of lasers is ablation of tissue together with effective hemostasis, minimal swelling and virtually no pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with the need for a single-tooth replacement in the maxilla by implant and simultaneous GBR

Exclusion Criteria:

* general contraindication for bone augmentation or implant surgeries,
* existence of swelling or pain at the time of surgery,
* smoking habits, pregnancy, and lactation.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
post-operative swelling intensity | Within the first 6 days after surgery
  Swelling on the operated side was evaluated as follows: 0 (none: no inflammation), 1 (mild: intraoral swelling confined to the surgical field), 2 (moderate: extra oral swelling in the surgical zone), or 3 (intense: extra oral swelling spreading beyond the surgical zone).

SECONDARY OUTCOMES:
post-operative pain intensity | Within the first 6 days after surgery
  Postoperative pain was measured using a visual analog scale (VAS) ranging from zero for "no pain" to 100 for "the worst possible pain".(questionnaire)
implant success | 3 months later
  based on Albrektsson success criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Tehran University of Medical Sciences, Tehran, Tehran Province
  - Neda Moslemi, Tehran, Tehran Province